CLINICAL TRIAL: NCT01548716
Title: A Cross-sectional Analysis of 25-hydroxy Vitamin d Levels in Non-itching Hemodialysis Patients
Brief Title: A Study of 25-hydroxy Vitamin d Levels in Non-itching Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Winthrop University Hospital (Other)
Collaborators: National Kidney Foundation, United States (Other)
Responsible Party: Principal Investigator, Mary Schanler, Administrative Dietitian, Winthrop University Hospital
Other Study IDs: 11318
Record Dates: First submitted 2012-02-24; First posted 2012-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Vitamin D Deficiency; End Stage Renal Disease
Keywords: Pruritis in hemodialysis patients; 25-Vitamin D in chronic kidney disease
MeSH Terms: conditions — Vitamin D Deficiency; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis:

25-hydroxy vitamin D levels in non-itching hemodialysis (HD) patients will be higher than those in HD patients with itching

25-hydroxy vitamin D levels will be measured in non-itching hemodialysis patients and compared to levels previously measured in a previous study of 25-hydroxy vitamin D levels of patients complaining of itching.

DETAILED DESCRIPTION:
25-hydroxy vitamin D levels from non-itching HD patients in this study will be compared to 25-hydroxy vitamin D levels from our ongoing study in HD patients with itching. The primary endpoints for both studies are continuous variables. Student's t test will be used to test for statistical significance. Multiple regression analysis will be used for controlling covariates and testing the interaction among covariates.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis treatment for > 3 months No complaints of itching within 1 month prior to study enrollment

Exclusion Criteria:

* Age < 18 years
* Failure to provide informed consent
* Intact PTH < 70 pg/ml or > 1,000 pg/ml
* Serum phosphorus > 7.0
* Serum calcium (adjusted for albumin)> 11
* Active malignancy
* Likelihood of imminent renal transplantation
* Current ergocalciferol treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients on hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
25 hydroxy vitamin D level | up to 2 weeks
  Pt will have blood sample taken and fill out 1) Pruritis Survey 2) Phosphorus Restriction Compliance Survey

CONTACTS AND LOCATIONS:
Overall Officials: Mary Schanler, RD, Principal Investigator — Winthrop University Hospital
Locations (2):
- United States (2):
  - Winthrop University Hospital Dialysis Unit, Mineola, New York
  - Winthrop University Hospital, Mineola, New York